CLINICAL TRIAL: NCT04386213
Title: A Prospective, Multicenter, Randomized Trial in Evaluating the Safety and Efficacy of the Paclitaxel Drug-coated Coronary Artery Balloon Catheter in Patients With Coronary Artery In-stent Restenosis Compared to SeQuent® Please Paclitaxel Drug-coated Coronary Artery Balloon Catheter
Brief Title: Trial for MicroPort's DCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROMISE-DCB
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery In-stent Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel Drug-coated Balloon (Experimental)
  Interventions: Device: coronary artery in-stent restenosis
- SeQuent® Please Paclitaxel Drug-coated Balloon (Active Comparator)
  Interventions: Device: coronary artery in-stent restenosis

INTERVENTIONS:
Device: coronary artery in-stent restenosis — treat the petients with coronary artery in-stent restenosis

SUMMARY:
This study is a multicenter, randomized, controlled clinical research and aims to evaluate the safety and efficacy of the paclitaxel drug-coated coronary artery balloon catheter in patients with coronary artery in-stent restenosis compared to seQuent® please paclitaxel drug-coated coronary artery balloon catheter.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized controlled clinical study is designed to enroll 216 subjects with in-stent restenosis and randomly assign them to the trial and control groups on a 1:1 basis.The experimental group was treated with paclitaxel drug-coated coronary artery balloon catheter, and the control group was treated with SeQuent ® Please paclitaxel balloon catheter, which has been marketed. In-segment late lumen loss 9 months after surgery was the main end point of the study. All subjects were followed up clinically at 1 month, 6 months, 9 months, 1 year and 2 years after the surgery, and were followed up with angiography at 9 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

1.18-75 years of age, males or non-pregnant females; 2.With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction; 3.Restenosis after the first stent implantation, and more than 90 days after the stent implantation; 4.Patients with indications for coronary artery bypass graft surgery; 5.To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

* Angiographic Inclusion Criteria:

  1. One or two target lesions;
  2. Restenosis in the stent (including bare stent, permanent coating and biodegradable coating) : Mehran I, II and III stenosis;The diameter of the reference vessel ranges from 2.0mm to 4.0mm, and the length ≤40mm;
  3. The original stent diameter stenosis before surgery must be ≥70% or ≥50% with local ischemia;
  4. There should be no more than two lesions requiring interventional treatment, and the distance between the two lesions must be >10mm.

Exclusion Criteria:

* General Exclusion Criteria:

  1. Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
  2. Severe congestive heart failure (NYHA III and above) ,or left ventricular ejection fraction <30% (ultrasound or left ventricular angiography);
  3. The unstable arrhythmia, such as high risk ventricular extrasystole and ventricular tachycardia;
  4. Blood test prompted platelet counts of less than 100x10E9/L or greater than 700x10E9/L, white blood cells than 3x10E9/L; which was judged to be clinically significant by the researchers;
  5. Preoperative renal function serum creatinine >2.0mg/DL; receiving hemodialysis;
  6. Subjects with bleeding tendency, antiplatelet preparation and anticoagulant treatment contraindications, subjects unable to receive antithrombotic treatment, or subjects unable to tolerate DAPT treatment for three months;
  7. Previous history of peptic ulcer or gastrointestinal bleeding within 6 months;
  8. Patients with cerebral vascular accident or transient ischemic attack (TIA) within the previous 6 months, or with permanent neurological defects that may lead to non-compliance with the protocol;
  9. Allergic to aspirin, heparin, contrast agent, polylactic acid polymer and paclitaxel;
  10. The life expectancy of the subjects is less than 12 months;
  11. The researcher judged that the subjects had poor compliance and could not complete the study as required;Or for other reasons that the researchers consider inappropriate;
  12. Subjects who are participating in any other clinical trial, or who have participated in clinical trials of other drugs or medical devices before being enrolled and have not reached the main study endpoint;
  13. Pregnant or breast-feeding female subjects (women who may be pregnant must undergo a pregnancy test 7 days prior to baseline surgery).
* Angiographic Exclusion Criteria:

  1. In-stent restenosis without successful predilatation;
  2. Stent restenosis of vein grafts;
  3. Bridge stent restenosis;
  4. All three vessels were diseased and needed revascularization;
  5. Vessel diameter of branch opening in bifurcation lesions ≥2.5mm;
  6. Complete occlusion of blood flow at TIMI level 0 (Mehran type IV stenosis);
  7. The lesion was located in the left trunk and within 2mm from the opening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
In-segment Late Lumen Loss | 9 months after coronary angiography
  In-segment Late Lumen Loss

SECONDARY OUTCOMES:
Device success | during the procedure
  defined as residual stenosis ≤30% and TIMI3 blood flow after drug-eluting balloon dilation.
Procedural success | Immediately after the index procedure
  Defined as target lesions with residual stenosis ≤30% and TIMI3 blood flow after any interventional treatment, without thrombus or dissection need interention.
Clinical success | At time of procedure up to 7 days in hospital
  Defined as the absence of device-related composite endpoint events during hospitalization (up to 7 days after surgery) on the basis of procedural success.
Device-oriented composite endpoints (Target Lesion Failure) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  TLF is defined as the composited endpoints of cardiac death, target vessel myocardial infarction and ischemia-driven target lesion revascularization.
Patient-oriented composite endpoint (PoCE) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Patient-oriented composite endpoint is defined as all cause death, all myocardial infarction, and any revascularization.
Death (Cardiac, Non-cardiac) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Defined as death due to the following causes. Acute myocardial infarction; cardiac perforation/cardiac tamponade; arrhythmia or abnormal conduction; death due to surgical complications, including bleeding, vascular repair, transfusion response, or coronary artery bypass surgery; anything that does not rule out death from cardiac causes.
  Non-cardiac death: defined as death from causes other than the above cardiac causes.
The number and rate of Myocardial Infarction (MI) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Attributable to target vessel (TV-MI), Not attributable to target vessel (NTV-MI)
The number and rate of Target Lesion Revascularization (TLR) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Ischemia-driven TLR (ID-TLR), Not ischemia-driven TLR (NID-TLR)
The number and rate of Target Vessel Revascularization (TVR) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Ischemia-driven TVR (ID-TVR), Not ischemia-driven TVR (NID-TVR)
The number and rate of Any Revascularization | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Ischemia-driven , Not ischemia-driven
The number and rate of Thrombosis (per ARC definition) | 1 month, 6 months, 9 months, 1 year and 2 years after index procedure
  Timing (acute, sub-acute, late and very late) Evidence (Definite and Probable)
In-segment angiography binary restenosis (ABR, %) | 9 months after index procedure
  Defined as the proportion of subjects with restenosis occurring in the target lesion segment and the diameter stenosis ≥50%.Quantitative coronary angiography analysis (QCA) calculation (1- 9 months after the operation of the original stent restenosis in-segment residual minimum lumen diameter / reference vessel diameter) ×100%

IPD SHARING:
Plan to Share IPD: Undecided